CLINICAL TRIAL: NCT00000314
Title: To Study Predictive Values of M-CPP and Fenfluramine in Cocaine Addicts
Brief Title: M-CPP and Fenfluramine in Cocaine Addicts - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: NIDA-09468-3; R01-09468-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — 1-(3-chlorophenyl)piperazine

INTERVENTIONS:
Drug: M-CPP

SUMMARY:
The purpose of this study is to evaluate predictive value of M-CPP and fenfluramine challenges for outcome.

ELIGIBILITY:
Please contact site for information.

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1994-09; Primary Completion 1999-08 (Actual); Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Drug use
Hospitalization, arrests, jail, employment, psychiataric symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Laure Buydens-Branchey, M.D., Principal Investigator — VA Medical Center
Locations (1):
- VA Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Derived] Ulmann G, Jouinot A, Tlemsani C, Curis E, Kousignian I, Neveux N, Durand JP, Goldwasser F, Cynober L, De Bandt JP. Lean Body Mass and Endocrine Status But Not Age Are Determinants of Resting Energy Expenditure in Patients with Non-Small Cell Lung Cancer. Ann Nutr Metab. 2019;75(4):223-230. doi: 10.1159/000504874. Epub 2019 Dec 19. PMID 31865308